CLINICAL TRIAL: NCT03337152
Title: Developing a Methodology to Assess 8-aminoquinoline Associated Haemolytic Risk in Females Heterozygous for G6PD in Endemic Populations
Brief Title: Assessing a Risk Model for G6PD Deficiency
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: study met study halting rules
Sponsor: PATH (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 856370-2
Record Dates: First submitted 2017-10-27; First posted 2017-11-08 (Actual); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2019-05

CONDITIONS: Malaria, Vivax; G6PD Deficiency
MeSH Terms: conditions — Malaria, Vivax; Glucosephosphate Dehydrogenase Deficiency | interventions — Primaquine; Chloroquine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two arms. 1a will receive primaquine for 14 days, and Arm 1b will receive chloroquine for 3 days and concomitant primaquine for 14 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1A: primaquine (Other): Twelve males hemizygous for wildtype G6PD, 12 females homozygous for wildtype G6PD, and 12 females heterozygous for G6PD deficiency will be randomized to arm 1A. Participants in arm 1A will receive primaquine for 14 days at 0.5 mg/Kg. Drug administration will be directly observed.
  Interventions: Drug: primaquine
- 1B: chloroquine + primaquine (Other): Twelve males hemizygous for wildtype G6PD, 12 females homozygous for wildtype G6PD, and 12 females heterozygous for G6PD deficiency will be randomized to arm 1B. Participants will receive chloroquine for 3 days concomitant with primaquine for 14 days at 0.5 mg/Kg. Drug administration will be directly observed.
  Interventions: Drug: chloroquine + primaquine

INTERVENTIONS:
Drug: primaquine — Participants receive primaquine for 14 days at 0.5 mg/Kg. Drug administration will be directly observed.
  Arms: 1A: primaquine
Drug: chloroquine + primaquine — Participants will receive chloroquine for 3 days concomitant with primaquine for 14 days at 0.5 mg/Kg. Drug administration will be directly observed.
  Arms: 1B: chloroquine + primaquine

SUMMARY:
A clinical study designed to develop and inform an individual risk of hemolysis model based on individual red blood cell G6PD levels. Volunteers who are eligible to treatment with primaquine as per national guidelines and with confirmed normal G6PD levels as per the fluorescent spot test will be exposed to treatment regimens of either primaquine alone for 14 days or 3 day chloroquine with concomitant primaquine for 14 days. The volunteers will be followed intensively during treatment and for 14 days after treatment for haematologic measures, G6PD quantification, and drug level assays.

DETAILED DESCRIPTION:
Open label, randomized trial with 72 total participants assigned to one of two treatment arms. Each arm will have 36 participants comprised of 12 males hemizygous for wildtype G6PD, 12 females homozygous for wildtype G6PD, and 12 females heterozygous for G6PD with a normal fluorescent spot test (FST) (G6PD genotype abnormal with G6PD activity ≥40% and ≤80% of normal). Arm 1a will receive primaquine for 14 days, and Arm 1b will receive chloroquine for 3 days and concomitant primaquine for 14 days. All participants will be healthy volunteers without severe G6PD deficiency who will be followed for two weeks after completing their study drug dosing. Pregnant women and those breastfeeding will be excluded. Venous blood samples will be taken at regular intervals for haematologic measures, G6PD quantification, and drug level assays. G6PD levels will be measured both by spectrophotometry to provide whole blood G6PD levels normalized for hemoglobin, as well by flow cytometry to to provide red blood cell G6PD distributions throughout the treatment and post treatment. Changes in the G6PD distributions will be modeled, incorporating other critical haematological indicators collected throughout the study too.

ELIGIBILITY:
Inclusion Criteria:

* Previous G6PD test at Shoklo Malaria Research Unit (SMRU) clinic with one of following results: 1) G6PD homozygous wildtype females (G6PD genotype normal) 2) G6PD heterozygous females with a normal FST (G6PD genotype abnormal with G6PD activity ≥40% and ≤80% of normal ) 3) G6PD hemizygous wildtype males (G6PD genotype normal)
* Willing to participate and sign informed consent form
* Willing to allow donated samples to be used in future research
* Aged ≥18 years
* Ability (in the investigators' opinion) and willing to comply with all study requirements

Exclusion Criteria:

All participants:

* Malaria or other illness
* Recent history (within 20 days) of anti-malarial treatment
* History of allergy or adverse reaction to chloroquine or primaquine
* Blood transfusion in the past 3 months
* G6PD activity less than 40% normal activity or 3.00 IU/gHb by the quantitative G6PD spectrophotometric assay
* Haemoglobin ≤10 g/dL
* Presence of any condition which in the judgment of the investigator would place the subject at undue risk or interfere with the results of the study

Female participants only:

* Pregnancy at the time of screening
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Nosten, MD, PhD, Principal Investigator — Shoklo Malaria Research Unit (SMRU), Mahidol-Oxford Tropical Medicine Research Unit
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing plan will be completed by the time of completion of the study

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants were enrolled into the trial but had not been randomized at the time of the study halt. Those 6 participants were thus never assigned to a study group.
Groups:
- 1A: Primaquine: primaquine: Participants receive primaquine for 14 days at 0.5 mg/Kg.
- 1B: Chloroquine + Primaquine: chloroquine + primaquine: Participants will receive chloroquine for 3 days concomitant with primaquine for 14 days at 0.5 mg/Kg.
Period: Overall Study
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Started | 24 | 24
Completed | 13 | 13
Not Completed | 11 | 11
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Stopped drug dosing due to study halt | 6 | 7

BASELINE CHARACTERISTICS:
Population: Participants randomized to a treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Median (Full Range); unit: years] | 33.5 [19 to 63] | 38.5 [19 to 64] | 36 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Thailand | 24 | 24 | 48
G6PD Status [Count of Participants; unit: Participants] — G6PD deficiency status based on genotyping
  Participants
    Heterozygous Female | 5 | 4 | 9
    Homozygous Female | 11 | 12 | 23
    Hemizygous Male | 8 | 8 | 16
Hemoglobin [Median (Full Range); unit: g/dL] | 13.2 [10.1 to 17.1] | 12.65 [9.6 to 15.7] | 12.9 [9.6 to 17.1]
G6PD Concentration [Median (Full Range); unit: IU/g Hb] — Based on spectrometer measurement
  IU/g Hb | 7.66 [2.94 to 11.08] | 7.515 [3.55 to 12.66] | 7.58 [2.94 to 12.66]

OUTCOME MEASURES:

1. Primary Outcome: Change in Haemoglobin
Description: The change in haemoglobin from baseline on exposure to primaquine for P.vivax treatment over treatment course to hemoglobin level at day 28.
Time Frame: 28 days after enrollment
Population: Among those with available data at baseline and at least one timepoint after study treatment began.
Measure: Median (Full Range); unit: g/dL
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 24 | 24
g/dL | -1.1 [-4.1 to 0] | -1.05 [-4.5 to 0]

2. Primary Outcome: Change in G6PD Concentration
Description: The haemoglobin-related change in G6PD concentration, as determined by spectrometer, over treatment course.
  Change is determined from baseline to day 28
Time Frame: 28 days after enrollment
Population: Among those with available data at baseline and at least one timepoint after study treatment began.
Measure: Median (Full Range); unit: IU/g Hb
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 24 | 24
IU/g Hb | -1.23 [-2.99 to -0.34] | -1.94 [-6.09 to -0.39]

3. Secondary Outcome: Significance of CYP2D6
Description: relevance of Dextromethorphan assay results to risk of haemolysis models
Time Frame: 28 days after enrollment
Population: Analysis not possible due to the study termination as the planned risk model could not be developed without sufficient data. Relevance of CYP2D6 results in the model thus unable to be determined.
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Association of Drug Levels
Description: Association of chloroquine and primaquine drug levels at the time of sampling for haematological and G6PD profiles.
Time Frame: Days 1,2,3,5,7,9,11,14,17,21
Population: This association was dependent on developing a model which requires completion of the study for an appropriate sample size. The incompletion of the study resulted in it not being possible to generate this model and therefore assess the association of drug levels with hematological and G6PD activity levels
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serious Adverse Events
Description: frequency of serious adverse events in women heterozygous for G6PD
Time Frame: 28 days after enrollment
Population: All randomized women heterozygous for G6PD.
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 5 | 4
Participants | 3 | 1

6. Secondary Outcome: Significance of Reticulocyte Count
Description: relevance of reticulocyte count to risk of haemolysis models
Time Frame: Days 1,2,3,5,7,9,11,14,17,21
Population: The relevance of reticulocyte count was dependent on developing a model which requires completion of the study for an appropriate sample size. The incompletion of the study resulted in it not being possible to generate this model and therefore assess the relevance of reticulocyte count on risk of hemolysis
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Significance of Urobilinogen Levels
Description: relevance of urobilinogen tests to risk of haemolysis models
Time Frame: Days 1,2,3,5,7,9,11,14,17,21
Population: The relevance of urobilinogen tests of was dependent on developing a model which requires completion of the study for an appropriate sample size. The incompletion of the study resulted in it not being possible to generate this model and therefore assess the relevance of urobilinogen tests on hemolytic risk models
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days after enrollment
Arm/Group | 1A: Primaquine | 1B: Chloroquine + Primaquine
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24 | 1/24
Other Adverse Events (participants affected / at risk) | 8/24 | 17/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Primaquine (N=24) | 1B: Chloroquine + Primaquine (N=24)
Hemolysis (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — Drug-induced anemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Primaquine (N=24) | 1B: Chloroquine + Primaquine (N=24)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 6 (6)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Decreased appetite (Gastrointestinal disorders) | 2 (2) | 5 (6)
Difficulty sleeping (General disorders) | 2 (2) | 5 (5)
Dizziness (General disorders) | 1 (1) | 11 (12)
Fatigue (General disorders) | 2 (2) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glucosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 4 (4) | 3 (3)
Methemoglobinemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Viral infection (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Elevated liver function test (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study met study halting rules and was terminated early. As a result, the full sample size was not enrolled and a complete data set was not available. Thus, the objectives of assessing and developing a G6PD risk model could not be met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT03337152/Prot_SAP_000.pdf